CLINICAL TRIAL: NCT00031395
Title: Clonidine in Attention Deficit Hyperactivity Disorder (ADHD) Treatment (CAT)
Brief Title: Clonidine in Attention Deficit Hyperactivity Disorder (ADHD) in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Floyd R. Sallee, M.D., Ph.D., Professor, University of Cincinnati School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS039087 (NIH)
Record Dates: First submitted 2002-03-04; First posted 2002-03-05 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; clonidine; methylphenidate; MPH
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Clonidine; Methylphenidate; 5,10-dihydro-5-methylphenazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator)
  Interventions: Drug: clonidine
- 2 (Active Comparator)
  Interventions: Drug: methylphenidate
- 3 (Active Comparator)
  Interventions: Drug: clonidine; Drug: methylphenidate
- 4 (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: clonidine — Clonidine is FDA-approved for the treatment of hypertension in adults.
  Arms: 1; 3
Drug: methylphenidate — MPH is FDA-approved for the treatment of ADHD symptoms in children.
  Other Names: MPH
  Arms: 2; 3
Other: placebo — an inactive substance
  Arms: 4

SUMMARY:
The purpose of this study is to determine the safety and efficacy of clonidine alone or in combination with methylphenidate for children 7-12 years of age with attention-deficit, hyperactivity disorder.

DETAILED DESCRIPTION:
This trial will compare the benefits and side effects of two medications-clonidine and methylphenidate (MPH)-used alone or in combination to treat ADHD in children. MPH is FDA-approved for the treatment of ADHD symptoms in children, and clonidine is FDA-approved for the treatment of hypertension in adults. Stimulant medications such as MPH are known to be safe and effective for the treatment of many ADHD symptoms. Such medicines, however, do not cure the condition or improve all of the symptoms of ADHD, and the long-term effectiveness of these medications is not well-known. In this study the participants will be randomly selected to receive one of four treatments: 1.) clonidine; 2.) MPH; 3.) clonidine and MPH; or 4.) a placebo (which is not an active medication, but a substance that is thought to have no biological effect). The time participation in the study is 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 through 12 in school.
* All subjects must meet DSM IV criteria for the diagnosis of ADHD of any subtype [21].
* Each subject must also satisfy the following criteria regarding the severity of ADHD symptoms: 1. ADHD must be viewed as clinically significant and worthy of treatment by medications as judged by the parent and the site investigator. Operationally, medication treatment will be considered indicated for any subject who has ADHD symptoms that significantly interfere with academic or social functioning and that have not improved (or are not expected to improve) sufficiently with non-pharmacological interventions (e.g., modifying the classroom environment, tutoring). 2. The site investigator's rating of global functioning on the C-GAS must yield a score of 70 or below. Scores below 70 on the C-GAS are designated as indicating abnormal function [22]. The score of 70 corresponds to the anchor point description: "Some difficulty in a single area, but generally functioning pretty well."
* Screen of Intelligence using the vocabulary and block design subtests of the Wechsler Intelligence Scale for Children-Third Edition indicates an estimated I.Q > 70.
* Informed consent/assent signed. We will not enroll any child who does not want to participate.
* The designated school for each subject agrees to participate in the study by completing all required questionnaires and following all specified procedures.
* The child must be able to swallow the tablets and capsules used in this study.

Exclusion Criteria:

* Subjects with tic disorder of any type or tic symptoms, a primary diagnosis of major depression, pervasive developmental disorder, autism, any psychotic disorder, and mental retardation (based on current DSM criteria) will be excluded. We will not exclude subjects with obsessive-compulsive disorder, oppositional-defiant disorder or conduct disorder.
* The presence of a known medical condition that would preclude the use of MPH or clonidine.
* Known pregnancy. A urinary pregnancy test will be performed for all menstruating female subjects. Female subjects of child bearing potential will be advised not to become pregnant. In this circumstance, study medication will be tapered and discontinued and the subject will be terminated from the study. A urinary pregnancy test will be repeated at the end of the study. Subjects who request information regarding possible birth control mechanisms will be referred to their primary care physicians.
* Known presence of impaired renal function. A routine urinalysis will be performed for each subject to exclude signs of renal failure.
* Known active cardiovascular disease/anomaly, which would be a contraindication for the use of MPH or clonidine.
* Subjects may not receive any other medication for the treatment of ADHD. Treatment with MPH or other stimulants must be discontinued for at least 2 weeks prior to enrollment and treatment with other medications to treat ADHD (e.g., antidepressants, clonidine) must be discontinued for at least 6 weeks prior to enrollment.
* Subjects may not receive any other psychotropic medication (e.g., serotonin reuptake inhibitors), anxiolytics (e.g., clonazepam) or hypnotics. Any such medication must be discontinued at least 6 weeks prior to enrollment.
* Previous use of MPH or clonidine will be permitted.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 1999-09; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Efficacy outcome was change in score on the Conners Abbreviated Symptom Questionnaire for Teachers (ASQ-T) | at 16 weeks

SECONDARY OUTCOMES:
the ASQ-Parent (ASQ-P) and Child Global Assessment Scales (C-GAS). Adverse events were monitored using AE logs, the Pittsburgh Side Effects Rating Scale, vital signs and electrocardiograms | at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Floyd R. Sallee, M.D., Ph.D., Principal Investigator — Children's Hospital & Medical Center
Locations (4):
- United States (4):
  - SUNY Buffalo, Center For Children & Families, Buffalo, New York
  - University of Rochester, Department of Neurology, Rochester, New York
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Cannon M, Pelham WH, Sallee FR, Palumbo DR, Bukstein O, Daviss WB. Effects of clonidine and methylphenidate on family quality of life in attention-deficit/hyperactivity disorder. J Child Adolesc Psychopharmacol. 2009 Oct;19(5):511-7. doi: 10.1089/cap.2009.0008. PMID 19877975